CLINICAL TRIAL: NCT00610090
Title: A Phase II, Single-arm, Prospective Study of the Safety of the UniFit Aorto-uni-iliac Endoluminal Stent Graft for the Repair of Abdominal Aortic Aneurysms
Brief Title: Safety Study for the Treatment of Abdominal Aortic Aneurysms
Acronym: UNITE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Duke Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMV-AUI-P2-001
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-05

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: UNITE; AAA; Abdominal Aortic Aneurysms; Stent; Graft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment - UniFit AAA Stent Graft (Experimental)
  Interventions: Device: UniFit AAA Stent Graft

INTERVENTIONS:
Device: UniFit AAA Stent Graft — Endovascular repair of Abdominal Aortic Aneurysms
  Other Names: UniFit; Unite Trial

SUMMARY:
The primary study objective, at this time, is to follow out to 5 years post implant the safety of already enrolled subjects who were treated with the UniFit Aorto-uni-iliac (AUI) Endoluminal Stent Graft (the "study device") for the repair of abdominal aortic aneurysms (AAAs).

DETAILED DESCRIPTION:
This is a phase II, single-arm, prospective study of the safety of the study device for the repair of AAAs.

The investigator will identify eligible patients and explain the study and study device placement procedure to each patient and/or any available family members. Patients who provide written informed consent will be evaluated for study eligibility within the time period identified under Duration of Treatment. Patients who are confirmed to be eligible, based on screening assessment findings, will be enrolled in the study.

After hospital discharge, patients will attend study center visits at 30 days, 6 months, and 1, 2, 3, 4, and 5 years post-procedure for follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has a AAA that meets one of the following criteria:

  1. Aneurysm diameter of greater than 4.5 cm, or less than 4.5 cm with rapid expansion
  2. The aneurysm has a saccular configuration where potential for rupture is increased or has exhibited dissection with potential for rupture at, or compromised flow to, vital structures
* The vessels immediately proximal and distal to the lesion are capable of accommodating the study device
* The access artery diameter and profile of the artery are capable of study device delivery.
* Patient has proximal and distal neck lengths of greater than or equal to 1.0 cm
* Patient is willing and able to comply with the follow-up regime.
* Patient has provided written informed consent.

Exclusion Criteria:

* Patient has an aortic diameter greater than 36 mm.
* Patients with ASA score less than 3 and deemed low risk by the Investigator for open surgical repair.
* Patient has an indispensable inferior mesenteric artery.
* Patient has a distal landing zone of < 2 cm in length or > 16 mm in diameter
* Patient has iliac arteries whose tortuosity prevents passage of the introducer catheter.
* If female, patient is pregnant
* Patient has a life expectancy less than two years.
* Patient has an allergy to any of the study device materials
* Patient has coagulopathy or bleeding disorders
* Patient for whom contrast medium or anticoagulation drugs are contraindicated
* Patient has an uncontained rupture of the aneurysm.
* Patient has an active systemic or localized groin infection
* Patient has a connective tissue disease.
* Patient has a GFR < 30 ml/min/1.73m2
* Patient has a circumferential mural thrombus at the implantation site.
* Patient is a candidate for a bifurcated endovascular graft.
* Patient has an aortic trunk with an angle greater than 90°.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 5 year
  The primary objective, at this time, is to ensure the safety of already enrolled and treated subjects. The data resulting from this study will not be used for any regulatory or commercialization purpose.
  The current sponsor, Duke Vascular, Inc. is requesting closure of this IDE

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Loma Linda VA, Loma Linda, California
  - UCLA Medical Center, Torrance, California
  - Christiana Hospital, Newark, Delaware
  - Florida Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Emory University, Atlanta, Georgia
  - Savannah Vascular Institute, Savannah, Georgia
  - Indiana University Hospital, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Englewood Hospital, Englewood, New Jersey
  - Albany Medical Center Hospital, Albany, New York
  - Dotter Interventional Institute, Portland, Oregon
  - Scott and White Hospital, Temple, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Sentara Healthcare, Vascular and Transplant Specialists, Norfolk, Virginia
  - Southwest Washington Medical Center, Vancouver, Washington